CLINICAL TRIAL: NCT03888573
Title: Which is Better to Decompress the Nerve Roots in Cervical Radiculopathy: Stretching or Traction From Foraminal Opening Position
Brief Title: Stretching Versus Traction in Patients With Cervical Radiculopathy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Farag Hanafy, Lecturer of Biomechanics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: nerve root decompression
Record Dates: First submitted 2019-03-20; First posted 2019-03-25 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Cervical Radiculopathy
Keywords: Stretching, Traction Decompression
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned into two groups; A and B. Patients within Group (A) will receive stretching protocols to the cervical musculature at the side of symptoms. Group (B) will be treated with traction from 15-degree flexion, 30-degree lateral bending, and 15-degree rotation toward the painful side.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stretch (Active Comparator): Patients within Stretch Group will receive stretching protocols to the cervical musculature at the side of symptoms.
  Interventions: Other: Stretching protocol
- Traction (Active Comparator): Patients within Traction Group will be treated with traction from 15-degree flexion, 30-degree lateral bending, and 15-degree rotation toward the painful side.
  Interventions: Other: Stretching protocol

INTERVENTIONS:
Other: Stretching protocol — Patients within Stretch Group will receive stretching protocols to the cervical musculature at the side of symptoms. Traction Group will be treated with traction from 15-degree flexion, 30-degree lateral bending, and 15-degree rotation toward the painful side.
  Other Names: Traction using The Triton decompression system

SUMMARY:
The purpose of the study is to compare the effects of traction decompression and neck muscle stretching on the magnitude of Flexor Carpi Radialis H-Reflex(HR), Neck Disability Index (NDI), and Visual Analogue Scale (VAS) pain scores in patients with cervical radiculopathy.

DETAILED DESCRIPTION:
Cervical traction has long been used to relieve compression of nerve roots caused by intervertebral discs. Yet, there is lack of knowledge that compares the effect of traction decompression with neck muscles stretching in patients with cervical radiculopathy

ELIGIBILITY:
Inclusion Criteria:

* Patients should have C5-C6 and C6-C7 paramedian disc protrusion manifested by unilateral symptoms in C6-C7 roots dermatome and myotomes of the upper extremities.
* They were diagnosed as cervical disc protrusion (C5- C7) for at least three months.
* All patients should have a second grade of disc bulge (2-3mm) which was detected from T2 axial view of MRI.

Exclusion Criteria:

* Patients will be excluded from the study if they have upper cervical spine disc pathology, cord compression and upper motor neuron symptoms, curvature abnormalities of the neck including reversed curve (kyphotic) and deformities, cervical rib syndrome, double crush syndrome, diabetic neuropathy, text neck , short neck (Churchill neck), Marked facet joint, neuro-central joint arthropathic pathology, osteoporosis.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
The Flexor Carpi radialis H-reflex | change from Baseline after 6-week of treament
  The peak-to-peak amplitudes of the four FCR-HR traces will be measured and averaged for each patient

SECONDARY OUTCOMES:
The Visual Analogue Scale Pain Scores(VAS) | Change from Baseline after 6-week of treament
  A 10-cm VAS was used for assessing pain intensity. It is a line whose ends are labeled as the extremes of pain; no pain and very extreme pain. The line is marked at intervals 1 cm each without any label. Patients will be simply asked to indicate which point along the line that best represents the intensity of perceived pain. The distance from the "no pain" end to the mark made by the patient will be measured as the patient's pain intensity score.
The Neck Disability Index (NDI) | Change from Baseline after 6-week of treatment
  The NDI will be measured on a 6-point scale from 0 (no disability) to 5 (full disability). The numeric response for each item will be summed for a score varying from 0 to 50. The NDI consists of 10 sections, each section the total possible score is 5, if the first statement is marked; the section score = 0, if the last statement is marked it = 5. The patients will choose the best choice that reflect his current state. If all ten sections are completed the score is calculated by dividing the obtained score on the total number of scores e.g. if the score recorded by the patients was (40) so the NDI=(40/50)x100=80%

CONTACTS AND LOCATIONS:
Overall Officials: Samiha Hafez Hassan, Prof., Study Chair — Professor of Physical Therapy for Neurology, Department of Physical Therapy for Neuromuscular Disorder and its Surgery, Faculty of Physical Therapy, Cairo University.; Salam Mohamed Elhafez, Prof., Study Director — Professor and Head of Department of Biomechanics, Faculty of Physical Therapy, Cairo University, Egypt.

REFERENCES:
- [Background] Caridi JM, Pumberger M, Hughes AP. Cervical radiculopathy: a review. HSS J. 2011 Oct;7(3):265-72. doi: 10.1007/s11420-011-9218-z. Epub 2011 Sep 9. PMID 23024624
- [Background] Graham N, Gross A, Goldsmith CH, Klaber Moffett J, Haines T, Burnie SJ, Peloso PM. Mechanical traction for neck pain with or without radiculopathy. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD006408. doi: 10.1002/14651858.CD006408.pub2. PMID 18646151